CLINICAL TRIAL: NCT00262444
Title: Effectivity and Efficiency of Turning Frequencies: a Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Distrac (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2003/084
Record Dates: First submitted 2005-12-04; First posted 2005-12-06 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Pressure Ulcer Lesions (Grade 2 or More)
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Different turning frequencies

SUMMARY:
Evaluation of the difference in pressure ulcer incidence or the time to develop pressure ulcers depending on the turning frequencies.

DETAILED DESCRIPTION:
Evaluation of the difference in pressure ulcer incidence or the time to develop pressure ulcers depending on the turning frequencies.

ELIGIBILITY:
Inclusion Criteria:

* non-blanchable erythema above a bony prominence
* Informed consent

Exclusion Criteria:

* Pressure ulcers grade 3 or 4
* Turning contra-indicated based on medical grounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2003-09; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Incidence of pressure ulcers | during 5 weeks
Time to develop pressure ulcers

SECONDARY OUTCOMES:
Different risk factors: age, length, weight, incontinence, urinary catheter, blood pressure, mobility, activity, diabetes, CVA, KATZ score, medication, duration in a sitting posture

CONTACTS AND LOCATIONS:
Overall Officials: Tom Defloor, PhD, Principal Investigator — University Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Result] Vanderwee K, Grypdonck MH, De Bacquer D, Defloor T. Effectiveness of turning with unequal time intervals on the incidence of pressure ulcer lesions. J Adv Nurs. 2007 Jan;57(1):59-68. doi: 10.1111/j.1365-2648.2006.04060.x. PMID 17184374
- See also: Website of the University Ghent — http://www.ugent.be